CLINICAL TRIAL: NCT04290884
Title: The Use of Tranexamic Acid in Chinese Elderly Patients Undergoing Femoral Nailing for Intertrochanteric Fracture: A Randomized Controlled Trial
Brief Title: Tranexamic Acid in Chinese Elderly Patients With Intertrochanteric Fracture RCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Wong Tak-Man, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UW 18-038
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Fracture of Femur
Keywords: elderly; intertrochanteric fracture
MeSH Terms: conditions — Femoral Fractures; Hip Fractures | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Local administration of tranexamic acid (Experimental): 1. All patients hip fracture will be treated according to the hospital standard procedure
  2. Check complete blood count on admission and Day 3 post-operation.
  3. 10ml tranexamic acid injected under the deep fascia around the fracture site under x-ray control
  4. Sealed envelope system: Operation room nurse will open a sealed envelope for treatment allocation. The medications are prepared by the nurse according to the instruction inside the envelop.
  5. Transfusion when clinically indicated or Hb < 8g/dL
  6. Blood Loss calculation (formula of Nadler, Hidalgo and Bloch)
  7. Blood taken at Day 3 post-operation will be used for measure of postoperative haematocrit. By this time postoperatively fluid shift has settled and the patient is haemodynamically stable.
  8. After discharge, patients will be seen in 6 weeks and 3 months
  Interventions: Drug: Tranexamic Acid
- Control group (No Intervention): 1. All patients hip fracture will be treated according to the hospital standard procedure
  2. Check complete blood count on admission and Day 3 post-operation.
  3. 10ml normal saline injected under the deep fascia around the fracture site under x-ray control
  4. Sealed envelope system: Operation room nurse will open a sealed envelope for treatment allocation. The medications are prepared by the nurse according to the instruction inside the envelop.
  5. Transfusion when clinically indicated or Hb < 8g/dL
  6. Blood Loss calculation (formula of Nadler, Hidalgo and Bloch)
  7. Blood taken at Day 3 post-operation will be used for measure of postoperative haematocrit. By this time postoperatively fluid shift has settled and the patient is haemodynamically stable.
  8. After discharge, patients will be seen in 6 weeks and 3 months

INTERVENTIONS:
Drug: Tranexamic Acid — The recruited patients will be randomly assigned to two groups, 50% chance to the experimental group (use of tranexamic acid) and 50% chance to the control group (use of normal saline). After the reduction of the intertrochanteric fracture, 10ml of tranexamic acid is injected under the deep fascia around the fracture area before inserting a drain. As for the control group, 10ml of normal saline is injected instead. Blood will be taken on the third day post operation, and the patient will be seen at 6 weeks, and 3 months.
  Other Names: Transamin
  Arms: Local administration of tranexamic acid

SUMMARY:
Hip fracture posed a major challenge to the health care system, with the one-year mortality of hip fracture reported as being approximately 20%. Perioperative haemoglobin level was associated with functional level of the patient and even mortality.

Different methods for administration of tranexamic acid had been described. It was well established that systemic administration of tranexamic acid could reduce perioperative blood loss and transfusion rate. Topical administration had been shown to decrease blood loss and transfusion rate.

The objective of our study is to investigate the hypothesis that tranexamic acid will reduce blood loss and transfusion rate in elderly patients undergoing hip fracture surgery.

DETAILED DESCRIPTION:
The incidence of geriatric hip fractures is projected to increase by more than 250% in the next twenty-five years as the world population ages. Hip fracture in elderly patients are associated with significant morbidity and mortality. One of the significant morbidity is blood loss, which has been reported as high as 1500ml. Blood loss may lead subsequent blood transfusion. The rate of blood transfusion has been reported between 20 to 60%. Blood loss and subsequent blood transfusion could lengthen the overall hospital length of stay and delay the rehabilitation.

Tranexamic acid, one of antifibrinolytic agents, is a synthetic derivative of the amino acid lysine and acts as a competitive inhibitor in the activation of plasminogen to plasmin, therefore preventing the degradation of fibrin. Shakur et al. reported that the use could reduce mortality in trauma patients. Tranexamic acid has been widely used in elective orthopaedic surgery such as total joint replacement and spine surgery. Several authors reported that tranexamic acid could decreases the blood loss, transfusion rate and cost.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 60
* Acute isolated intertrochanteric fracture and sub trochanteric fracture treated with short proximal femoral nailing

Exclusion Criteria:

* Use of any anticoagulant at the time of admission
* Documented allergy to tranexamic acid
* History of pulmonary embolism or deep vein thrombosis
* Hepatic failure
* Severe renal insufficiency
* Active coronary artery disease in the past 12 months
* History of cerebrovascular accident in the past 12 months
* Presence of a drug-eluting stent
* Active oncological diseases
* Coagulopathy (international normalised ratio (INR)>1.4)
* Pathological fractures
* Periprosthetic fractures
* Operation >2 days from admission

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-05-23 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Transfusion rate | Day 3 post operation
  The total blood transfusion post operation
Blood loss | Day 3 post operation
  Blood loss calculation according to formula of Nadler, Hidalgo and Bloch

SECONDARY OUTCOMES:
3 months mortality rate | from post operation to 3 months
  mortality rate of the patient within post operation 3 months
Complications | from post operation to 3 months
  Complications related to thrombotic events

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schneider EL, Guralnik JM. The aging of America. Impact on health care costs. JAMA. 1990 May 2;263(17):2335-40. PMID 2109105
- [Background] Bhaskar D, Parker MJ. Haematological indices as surrogate markers of factors affecting mortality after hip fracture. Injury. 2011 Feb;42(2):178-82. doi: 10.1016/j.injury.2010.07.501. PMID 20850741
- [Background] Foss NB, Kristensen MT, Kehlet H. Anaemia impedes functional mobility after hip fracture surgery. Age Ageing. 2008 Mar;37(2):173-8. doi: 10.1093/ageing/afm161. PMID 18349013
- [Background] Lawrence VA, Silverstein JH, Cornell JE, Pederson T, Noveck H, Carson JL. Higher Hb level is associated with better early functional recovery after hip fracture repair. Transfusion. 2003 Dec;43(12):1717-22. doi: 10.1046/j.0041-1132.2003.00581.x. PMID 14641869
- [Background] Zhang P, He J, Fang Y, Chen P, Liang Y, Wang J. Efficacy and safety of intravenous tranexamic acid administration in patients undergoing hip fracture surgery for hemostasis: A meta-analysis. Medicine (Baltimore). 2017 May;96(21):e6940. doi: 10.1097/MD.0000000000006940. PMID 28538384
- [Background] Drakos A, Raoulis V, Karatzios K, Doxariotis N, Kontogeorgakos V, Malizos K, Varitimidis SE. Efficacy of Local Administration of Tranexamic Acid for Blood Salvage in Patients Undergoing Intertrochanteric Fracture Surgery. J Orthop Trauma. 2016 Aug;30(8):409-14. doi: 10.1097/BOT.0000000000000577. PMID 26978136
- [Background] Tengberg PT, Foss NB, Palm H, Kallemose T, Troelsen A. Tranexamic acid reduces blood loss in patients with extracapsular fractures of the hip: results of a randomised controlled trial. Bone Joint J. 2016 Jun;98-B(6):747-53. doi: 10.1302/0301-620X.98B6.36645. PMID 27235515